CLINICAL TRIAL: NCT05990452
Title: A Phase I/II First-in-human Study of 9MW2921 to Evaluate the Safety, Tolerability and Preliminary Efficacy of 9MW2921 in Patients With Advanced Solid Tumors
Brief Title: Phase I/II FIH Study of 9MW2921 in Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9MW2921-2023-CP101
Record Dates: First submitted 2023-07-31; First posted 2023-08-14 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 9MW2921 (Experimental)
  Interventions: Drug: 9MW2921

INTERVENTIONS:
Drug: 9MW2921 — All subjects will receive 9MW2921 by intravenous (IV) every 3 weeks.

SUMMARY:
This is an open-label, Phase I-II, first-in-human (FIH) study of 9MW2921 in patients with locally advanced or metastatic solid tumors refractory to all standard therapies. The objective of this study is to evaluate the safety, tolerability, PK, immunogenicity and Preliminary Antitumor Activity of 9MW2921.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75 years old, male or female, voluntarily agree to participate in the study and sign the Informed Consent Form (ICF).
2. ECOG PS is 0 or 1.
3. Subjects must have histologically confirmed advanced and/or metastatic malignancies for which failure of standard treatment or lack/intolerant of effective standard treatment.
4. Subjects must be able to provide fresh or ≥5 slides of unstained tumor tissue.
5. Survival expectation of at least 3 months.
6. At least one measurable lesion according to RECIST v1.1.
7. The organ function level must meet the protocol requirements.
8. Women and men of reproductive age must agree to use effective contraception from the date of signing the informed consent until 6 months after the last administration of 9MW2921, and women of reproductive age must have negative serum pregnancy test results within 7 days prior to administration.
9. Ability and willingness to understand visits, treatment, laboratory tests and other study procedures.

Exclusion Criteria:

1. History of other malignancy within 3 years.
2. Subjects with active central nervous system (CNS) metastasis or meningeal metastasis.
3. History of treatment with topoisomerase I inhibitors.
4. Anti-tumor therapy such as traditional Chinese medicine or immunomodulatory drugs within 14 days prior to the first dose of study drug, or radiotherapy, chemotherapy, biological agents, immunotherapy within the previous 21 days.
5. Adverse reactions related to previous treatments failed to recover to CTCAE 5.0 ≤1.
6. Had major surgery within 28 days before dosing, or has surgery plan during the study time (including the screening time).
7. Subjects with clinically significant cardiovascular disease within 6 months prior to the first dose of study drug.
8. Any other serious or uncontrolled disease that, in the opinion of the investigator, would make it inappropriate to participate in the trial or would interfere with the subject's compliance with the trial protocol.
9. Subjects with active chronic inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease) or history of bowel obstruction, gastrointestinal perforation.
10. Live vaccine was administered within 28 days prior to first dose, or has plan to receive any kind of live vaccine during this study.
11. High-dose systemic corticosteroid administration within 2 weeks prior to the first dose of study drug.
12. Subjects who were allergic to any composition of investigational drug.
13. Prior autologous or allogeneic organ transplantation (except corneal transplantation) or stem cell transplantation prior to the first dose of study drug.
14. Subjects participate in other clinical trials such as medicine or medical device and use them within 28 days before the first dose.
15. Has a history of substance abuse, alcohol or drug abuse, or psychiatric illness.
16. Women who are pregnant or breastfeeding.
17. Other conditions deemed ineligible for this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose Limited Toxicity (DLT) | 21 Days (first cycle)
  To determine the dose limiting toxicities (DLTs) of 9MW2921
Adverse Events and Serious Adverse Events | up to 2 years or intolerable toxicity, disease progression or death, patient withdrawal of informed consent, withdrawal from the study and so on
  Percentage of patients with adverse events (AEs) and serious adverse events (SAEs)
ORR | up to 2 years or intolerable toxicity, disease progression or death, patient withdrawal of informed consent, withdrawal from the study and so on
  Defined as the percentage of subjects who experience a best response of either CR or PR.

SECONDARY OUTCOMES:
PK Parameters: Cmax | 1 years
  Maximum concentration(Cmax)
PK Parameters: AUC | 1 years
  The area under the curve (AUC)
PK Parameters: t1/2 | 1 years
  The half life(t1/2)
Incidence of ADAs Against 9MW2921 | up to 2 years
  The incidence of ADAs against 9MW2921 during the study will be summarized
Progression free survival(PFS) according to RECIST 1.1 | up to 2 years or intolerable toxicity, disease progression or death, patient withdrawal of informed consent, withdrawal from the study and so on
  Time from the date of first infusion to the earliest date of documented disease progression per radiological evidence or death from any cause
Duration of Response (DoR) according to RECIST 1.1 | up to 2 years or intolerable toxicity, disease progression or death, patient withdrawal of informed consent, withdrawal from the study and so on
  Time from the date of the first complete response (CR) or partial response (PR) to the earliest date of disease progression or death from any cause. DOR is only defined for subjects who have best overall response of CR or PR.
Disease Control Rate (DCR) according to RECIST 1.1 | up to 2 years or intolerable toxicity, disease progression or death, patient withdrawal of informed consent, withdrawal from the study and so on
  Defined as the percentage of subjects who experience a best response of CR, PR or stable disease (SD).

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Jian, Professor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Centel, Shanghai, China

IPD SHARING:
Plan to Share IPD: No